CLINICAL TRIAL: NCT01881399
Title: Fluorescence Cholangiography Versus Conventional Intraoperative Cholangiography for Visualization of Biliary Tract Anatomy : a Prospective, Controlled Study
Brief Title: Fluorescence Versus Intraoperative Cholangiography in the Visualization of Biliary Tree Anatomy
Acronym: FLARIOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-004; 2012-A01664-39 (Other: ANSM France)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Cholelithiasis; Gallbladder Polyps
Keywords: Cholelithiasis; Gallbladder polyps; Fluorescence; Indocyanine green (ICG); Intraoperative cholangiography (IOC); da Vinci surgical system
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorescence/Virtual cholangiography/IOC (Experimental): Prior to cholecystectomy, patients will undergo:
  * Fluorescence cholangiography (visualization following up to a maximum of 0.5 mg/kg ICG - usually 10 ml of 0,5 mg/ml solution)
  * Virtual cholangiography (enhanced-reality) superimposed on fluorescence images
  * Conventional IOC (intraoperative cholangiography)
  Interventions: Device: Fluorescence cholangiography (da Vinci surgical system); Other: Virtual cholangiography; Procedure: Conventional IOC

INTERVENTIONS:
Device: Fluorescence cholangiography (da Vinci surgical system) — Patients will received IV injection of ICG intra-operatively, allowing surgeons to view bile ducts under fluorescence imaging using the da Vinci surgical system with fluorescence Imaging system.
  Other Names: da Vinci Si surgical system with da Vinci Fluorescence Imaging Vision System
Other: Virtual cholangiography — Images from virtual cholangiography will be superimposed in real time on images obtained with fluorescence.
Procedure: Conventional IOC — Patients will undergo conventional intraoperative cholangiography (with use of radio-opaque dye), allowing surgeons to view bile ducts under Rx imaging.

SUMMARY:
The burden of iatrogenic bile duct injury (BDI), the most feared complication of laparoscopic cholecystectomy (LC), is extremely high and the repercussions on the patient's outcomes may be severe ranging from intraoperative repair to liver transplant or patient's death. Different techniques have been proposed to prevent BDI.

Our hypothesis is that a fluorescence-based Imaging would allow visualization of the biliary tree anatomy as good as with the Intraoperative Cholangiogram with several main advantages:

1. ease of use
2. lack of invasiveness
3. absence of ionizing radiation to the patient and the operating staff
4. performed prior to any dissection (prior to "critical view of safety")

Capacity of enhanced-reality based on virtual cholangiography (computer treatment of MRI images) to guide biliary tree anatomy visualization will be also evaluated in this study.

The study requires a 2-month patient participation.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years old
* Symptomatic gallbladder lithiasis or gallbladder polyps
* Clinical, biological ou medical imaging history leading to suspicion of gallstones migration
* Absence of contra-indication to anesthesia and cholecystectomy procedure
* Ability to understand the study related information and to provide written informed consent
* Registered with the French social security regime

Non inclusion Criteria:

* Inability to give informed consent
* Acute Cholecystitis
* Contraindications to MRI exam (claustrophobia, implantable devices)
* Potential risk of allergic reactions to iodine-containing contrast agents, to indocyanine green or other fluorescent compounds
* Pregnancy or breast-feeding
* Exclusion period from other clinical trial
* Forfeit freedom from an administrative or legal obligation
* Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of a ICG-fluorescence guidance in visualizing the biliary anatomy and to compare accuracy to conventional intraoperative cholangiography | Intra-operatively
  Percentage of patients for whom fluorescence allows for cysticocholedochal junction with precision at least as good as intraoperative cholangiography (identification of anatomical details and information).
  Independent aposteriori evaluation performed by a radiologist/surgeon team.

SECONDARY OUTCOMES:
To evaluate the ability of fluorescence-based imaging in visualizing the biliary tree anatomy | Intra-operatively
  Percentage of patients for whom fluorescence-based imaging allows correct identification of biliary tree anatomy (anatomical variant, cystic duct stones, bile duct stones, dilated ducts)
To evaluate the ability of enhanced reality in visualizing the biliary anatomy intra-operatively, especially the cysticocholedochal junction | Intra-operatively
  Percentage of patients for whom enhanced reality allows correct identification of biliary tree anatomy,especially the cysticocholedochal junction
To evaluate time required for the visualization of biliary tree anatomy for each modality : fluorescence, enhanced reality, conventional intraoperative cholangiography | Intra-operatively
  Time required for fluorescence-based exam, enhanced reality visualization, conventional intraoperative cholangiography Conversion to costs (based on mean cost of OR minute)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pessaux, Pr, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Diana M, Soler L, Agnus V, D'Urso A, Vix M, Dallemagne B, Faucher V, Roy C, Mutter D, Marescaux J, Pessaux P. Prospective Evaluation of Precision Multimodal Gallbladder Surgery Navigation: Virtual Reality, Near-infrared Fluorescence, and X-ray-based Intraoperative Cholangiography. Ann Surg. 2017 Nov;266(5):890-897. doi: 10.1097/SLA.0000000000002400. PMID 28742709